CLINICAL TRIAL: NCT01878292
Title: A Double-Blind, Placebo-Controlled Evaluation of the Safety and Efficacy of Vilazodone in Adolescent Patients With Major Depressive Disorder
Brief Title: Safety and Efficacy of Vilazodone in Adolescent Patients With Major Depressive Disorder
Acronym: VLZ-MD-21
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Forest Laboratories (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VLZ-MD-21
Record Dates: First submitted 2013-06-11; First posted 2013-06-14 (Estimated); Results first posted 2019-12-24 (Actual); Last update posted 2019-12-24 (Actual); Status verified 2019-12

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Vilazodone Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Placebo (Placebo Comparator): Dose-matched placebo tablets, once per day, oral administration
  Interventions: Drug: Placebo
- Vilazodone 15 mg (Experimental): 15 mg vilazodone tablets, once per day, oral administration
  Interventions: Drug: Vilazodone
- vilazodone 30 mg (Experimental): 30 mg vilazodone tablets, once per day, oral administration
  Interventions: Drug: Vilazodone

INTERVENTIONS:
Drug: Placebo — Dose matched placebo tablets, once per day, oral administration.
  Arms: Placebo
Drug: Vilazodone — Vilazodone tablets, 15 mg per day, oral administration
  Other Names: Viibryd
  Arms: Vilazodone 15 mg
Drug: Vilazodone — Vilazodone tablets, 30 mg once per day, oral administration
  Other Names: Viibryd
  Arms: vilazodone 30 mg

SUMMARY:
The purpose of this study is to evaluate the efficacy, safety, and tolerability of vilazodone relative to placebo in adolescent outpatients (12-17) with major depressive disorder.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female outpatients between 12-17 years of age
* Primary diagnosis of major depressive disorder (MDD)
* Children's Depression Rating Scale-Revised (CDRS-R) score of 40 or greater
* Clinical Global Impressions-Severity (CGI-S) score of 4 or greater

Exclusion Criteria:

* Current (past 3 months) principal Diagnostic and Statistical Manual of Mental Disorders, 4th edition, Text Revision (DSM-IV-TR) based diagnosis of an axis disorder other than major depressive disorder (MDD) that is the primary focus of treatment.
* History of suicidal behavior, or requires precaution against suicide
* Not generally healthy medical condition
* Seizure disorder

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 529 (Actual)
Dates: Start 2013-07-11 (Actual); Primary Completion 2016-03-17 (Actual); Study Completion 2016-10-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chandran Prakash, Study Director — Allergan
Locations (52):
- United States (52):
  - Forest Investigative Site 073, Imperial, California
  - Forest Investigative Site 052, Los Angeles, California
  - Forest Investigative Site 023, Murrieta, California
  - Forest Investigative Site 004, Orange, California
  - Forest Investigative Site 037, San Diego, California
  - Forest Investigative Site 006, Washington D.C., District of Columbia
  - Forest Investigative Site 039, Gainesville, Florida
  - Forest Investigative Site 009, Jacksonville Beach, Florida
  - Forest Investigative Site 063, Miami, Florida
  - Forest Investigative Site 034, Oakland Park, Florida
  - Forest Investigative Site 016, Orlando, Florida
  - Forest Investigative Site 064, Orlando, Florida
  - Forest Investigative Site 014, Atlanta, Georgia
  - Forest Investigative Site 030, Roswell, Georgia
  - Forest Investigative Site 032, Libertyville, Illinois
  - Forest Investigative Site 048, Naperville, Illinois
  - Forest Investigative Site 051, Terre Haute, Indiana
  - Forest Investigative Site 013, Overland Park, Kansas
  - Forest Investigative Site 070, Lake Charles, Louisiana
  - Forest Investigative Site 050, Baltimore, Maryland
  - Forest Investigative Site 054, Baltimore, Maryland
  - Forest Investigative Site 049, Rockville, Maryland
  - Forest Investigative Site 026, Watertown, Massachusetts
  - Forest Investigative Site 024, Rochester Hills, Michigan
  - Forest Investigative Site 015, Creve Coeur, Missouri
  - Forest Investigative Site 055, Saint Charles, Missouri
  - Forest Investigative Site 072, St Louis, Missouri
  - Forest Investigative Site 066, Las Vegas, Nevada
  - Forest Investigative Site 007, Cherry Hill, New Jersey
  - Forest Investigative Site 071, Neptune City, New Jersey
  - Forest Investigative Site 008, Albuquerque, New Mexico
  - Forest Investigative Site 057, Rochester, New York
  - Forest Investigative Site 059, Durham, North Carolina
  - Forest Investigative Site 053, Avon Lake, Ohio
  - Forest Investigative Site 021, Canton, Ohio
  - Forest Investigative Site 012, Cincinnati, Ohio
  - Forest Investigative Site 029, Columbus, Ohio
  - Forest Investigative Site 018, Oklahoma City, Oklahoma
  - Forest Investigative Site 011, Oklahoma City, Oklahoma
  - Forest Investigative Site 065, Tulsa, Oklahoma
  - Forest Investigative Site 040, Philadelphia, Pennsylvania
  - Forest Investigative Site 074, Charleston, South Carolina
  - Forest Investigative Site 062, Memphis, Tennessee
  - Forest Investigative Site 001, Dallas, Texas
  - Forest Investigative Site 027, Houston, Texas
  - Forest Investigative Site 041, Plano, Texas
  - Forest Investigative Site 045, The Woodlands, Texas
  - Forest Investigative Site 019, Clinton, Utah
  - Forest Investigative Site 060, Richmond, Virginia
  - Forest Investigative Site 035, Bellevue, Washington
  - Forest Investigative Site 068, Bothell, Washington
  - Forest Investigative Site 022, Kirkland, Washington

REFERENCES:
- [Derived] Durgam S, Chen C, Migliore R, Prakash C, Edwards J, Findling RL. A Phase 3, Double-Blind, Randomized, Placebo-Controlled Study of Vilazodone in Adolescents with Major Depressive Disorder. Paediatr Drugs. 2018 Aug;20(4):353-363. doi: 10.1007/s40272-018-0290-4. PMID 29633166

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Randomization and treatment assignment were based on a randomization scheme prepared by Allergan Biostatistics prior to the start of the study
Period: Randomized
Arm/Group | Placebo | Vilazodone 15 mg | Vilazodone 30 mg
Started | 174 | 175 | 180
Completed | 171 | 175 | 180
Not Completed | 3 | 0 | 0
Not completed — Protocol Violation | 1 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 0
Period: Double-blind Treatment Period
Arm/Group | Placebo | Vilazodone 15 mg | Vilazodone 30 mg
Started | 171 | 175 | 180
Completed | 142 | 149 | 161
Not Completed | 29 | 26 | 19
Not completed — Other Reasons | 2 | 0 | 0
Not completed — Lost to Follow-up | 6 | 3 | 1
Not completed — Withdrawal by Subject | 9 | 7 | 8
Not completed — Protocol Violation | 3 | 4 | 2
Not completed — Lack of Efficacy | 5 | 3 | 0
Not completed — Adverse Event | 4 | 9 | 8
Period: Double-blind Down-Taper Period
Arm/Group | Placebo | Vilazodone 15 mg | Vilazodone 30 mg
Started | 127 | 140 | 146
Completed | 122 | 132 | 142
Not Completed | 5 | 8 | 4
Not completed — Withdrawal by Subject | 5 | 8 | 4

BASELINE CHARACTERISTICS:
Population: The Safety Population consisted of all patients in the Randomized Population who took at least 1 dose of double-blind investigational product.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Vilazodone 15 mg | Vilazodone 30 mg | Total
Number analyzed (Participants) | 171 | 175 | 180 | 526
Age, Continuous [Mean (Standard Deviation); unit: Years] | 14.9 (1.7) | 14.9 (1.6) | 14.6 (1.6) | 14.8 (1.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 103 | 103 | 107 | 313
  Male | 68 | 72 | 73 | 213
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 21 | 22 | 19 | 62
  Not Hispanic or Latino | 150 | 153 | 161 | 464
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: Participants]
  White | 110 | 115 | 121 | 346
  Black or African American | 45 | 48 | 49 | 142
  Asian | 6 | 3 | 0 | 9
  American Indian or Alaska Native | 2 | 2 | 4 | 8
  Native Hawaiian/Other Pacific Islander | 0 | 0 | 0 | 0
  Other | 8 | 7 | 6 | 21
Weight [Mean (Standard Deviation); unit: kg] | 71.87 (20.78) | 70.10 (20.65) | 70.89 (20.58) | 70.95 (20.64)
BMI [Mean (Standard Deviation); unit: kg/m2] | 25.97 (7.15) | 25.30 (6.86) | 25.66 (6.70) | 25.64 (6.89)

OUTCOME MEASURES:

1. Primary Outcome: Change in Children's Depression Rating Scale - Revised (CDRS-R) Total Score
Description: The Children's Depression Rating Scale-Revised (CDRS-R) total score ranges from 17 (minimal or no symptoms of depression) to 133 (indicative of depression) is a semi-structured, clinician-rated instrument designed for use with children and adolescents between the ages of 6 to 17 years of age and their caregivers. The CDRS-R evaluates the presence and severity of symptoms commonly associated with depression in childhood.
Time Frame: From Baseline to week 8
Population: The Intent-to-Treat (ITT) Population will consist of all patients in the Safety Population who had baseline and at least 1 postbaseline assessment of the Children's Depression Rating Scale-Revised (CDRS-R) total score.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Vilazodone 15 mg | Vilazodone 30 mg
Number analyzed (Participants) | 170 | 174 | 180
units on a scale | -22.48 (0.921) | -22.94 (0.904) | -24.22 (0.872)

2. Secondary Outcome: Change in Clinical Global Impressions-Severity (CGI-S) Score
Description: The Clinical Global Impressions-Severity (CGI-S) is a clinician-rated instrument used to rate the severity of the patient's current state of mental illness compared with the clinician's total experience with patients with major depressive disorder (MDD). The severity of the patient's MDD was rated on a scale from 1 to 7, with 1 indicating a normal state and 7 indicating a patient who is among the most extremely ill patients.
Time Frame: From Baseline to Week 8
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Vilazodone 15 mg | Vilazodone 30 mg
Number analyzed (Participants) | 170 | 174 | 180
units on a scale | -1.60 (0.094) | -1.82 (0.092) | -1.87 (0.089)

ADVERSE EVENTS:
Time Frame: Adverse event data was collected for up to 10 weeks, including approximately 1 week of screening, an 8-week double-blind treatment period, and a 1-week double-blind down-taper period.
Arm/Group | Placebo | Vilazodone 15 mg | Vilazodone 30 mg
All-Cause Mortality (participants affected / at risk) | 0/171 | 0/175 | 0/180
Serious Adverse Events (participants affected / at risk) | 1/171 | 2/175 | 3/180
Other Adverse Events (participants affected / at risk) | 63/171 | 81/175 | 97/180
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=171) | Vilazodone 15 mg (N=175) | Vilazodone 30 mg (N=180)
Intentional overdose (Injury, poisoning and procedural complications) | 0 | 0 | 1
Pilonidal cyst (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Suicidal ideation (Psychiatric disorders) | 1 | 0 | 1
Suicide attempt (Psychiatric disorders) | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 1 | 0
Mental status changes (Psychiatric disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=171) | Vilazodone 15 mg (N=175) | Vilazodone 30 mg (N=180)
Nausea (Gastrointestinal disorders) | 14 | 53 | 50
Abdominal pain upper (Gastrointestinal disorders) | 11 | 7 | 28
Vomiting (Gastrointestinal disorders) | 6 | 11 | 21
Diarrhoea (Gastrointestinal disorders) | 8 | 15 | 16
Nasopharyngitis (Infections and infestations) | 6 | 6 | 13
Headache (Nervous system disorders) | 28 | 25 | 30
Dizziness (Nervous system disorders) | 5 | 8 | 13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All data generated in this study are the property of the sponsor. An integrated clinical and statistical report will be prepared at the completion of the study. Publication of the results by the Investigator will be subject to mutual agreement between the Investigator and the sponsor and will follow sponsor's standard operating procedures on publications.